CLINICAL TRIAL: NCT04038957
Title: An Open-Label Positron Emission Tomography Study to Investigate the Effect of Adjunctive Administration of SEP-363856 on Brain Dopamine Synthesis Capacity Using 18F-DOPA in Adult Subjects With Schizophrenia
Brief Title: A Clinical Study to Investigate the Effect of an Investigational Drug as an Added Medication to an Antipsychotic, in Adults With Schizophrenia, as Measured Positron Emission Tomography (PET) Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-118; 2019-000568-65 (EudraCT Number)
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: This is a single-site, open-label, flexibly-dosed study
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-363856 (Experimental): SEP-363856 50mg, 75mg flexible dosing, dosed once daily
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 50mg, 75mg flexable dosing, dosed once daily capsule

SUMMARY:
A clinical study to investigate the effect of an investigational drug as an added medication to an antipsychotic, in adults with schizophrenia, as measured positron emission tomography (PET) imaging . This study is accepting male and female participants between 18 years old -45 years old who have been diagnosed with schizophrenia. This study will be conducted in 2 locations in the UK. The study will last approximately 14 months.

DETAILED DESCRIPTION:
This is a single-site, open-label, flexibly-dosed study evaluating the effect on brain dopamine synthesis capacity as measured by 18F-DOPA PET imaging of adjunctive open-label administration of SEP-363856 (50 to 75 mg/day) over 2 weeks in adults with schizophrenia. The study will consist of 3 periods: Screening (up to 28 days), Treatment (2 weeks), and a Follow-up visit

ELIGIBILITY:
Inclusion Criteria:

-1. Subject must give written informed consent and privacy authorization prior to participation in the study.

2. Subject must be willing and able to comply with the study procedures and visit schedule, including required minimum week in-clinic treatment period, and must be able to understand and follow verbal and written instructions

* Male or female subject between 18 to 45 years of age (inclusive) at the time of consent
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a primary diagnosis of schizophrenia as established by clinical interview (using the DSM-5 as a reference and confirmed using the Structured Clinical Interview for DSM-V Clinical Trials Version [SCID-CT]). The duration of the subject's illness whether treated or untreated must be ≥ 6 months.
* Subject must be on a stable dose of a single antipsychotic medication, dosed within the labeled dose-range, for a minimum of 3 weeks prior to the PET scan at the screening visit. Patients taking clozapine are not eligible to participate
* Subject must have a Clinical Global Impression-Severity (CGI-S) score ≥ 3 (mild or greater)
* Subject must have a Positive and Negative Syndrome Scale (PANSS) total score ≥ 70.
* . Subject's BMI must be at least 18 kg/m2 but no more than 35 kg/m2.
* Female subjects must have a negative serum pregnancy test at screening; as well as a negative urine pregnancy test prior to the PET scan on each day PET scans are performed, as well as prior to the MRI scan.

  1. Female subject of childbearing potential and male subject with female partner of childbearing potential must agree to use an acceptable form of birth control from at least 30 days prior to administration of the first dose of study drug, during the treatment period, and 60 days after completion or premature discontinuation from the study drug. Male subjects must also refrain from semen/sperm donation 30 days prior to administration of the first dose of study drug, during the treatment period, and 60 days after completion or premature discontinuation from the study drug.

     * Adequate contraception is defined as continuous use of either two barrier methods (eg, condom and spermicide or diaphragm with spermicide) or a hormonal contraceptive. Acceptable hormonal contraceptives include the following: a) contraceptive implant (such as Norplant®) implanted at least 90 days prior to screening; b) injectable contraception (such as meroxyprogesterone acetate injection) given at least 14 days prior to screening; or c) oral contraception taken as directed for at least 30 days prior to screening. In the Investigator's judgment, the subject will adhere to this requirement.
  2. . Female subjects who are of non-childbearing potential are not required to abide by birth control requirements.

     - Non-childbearing potential is defined as subject who is surgically sterile, has undergone tubal ligation, or is postmenopausal (defined as at least 12 months of spontaneous amenorrhea or between 6 and 12 months of spontaneous amenorrhea with follicle stimulating hormone [FSH] concentrations within postmenopausal range as determined by laboratory analysis).
* Subject is, in the opinion of the Investigator, generally healthy based on screening medical history, PE, neurological examination, vital signs, clinical laboratory values (hematology, serum chemistry urinalysis, lipid panel, coagulation panel, thyroid panel, and serum prolactin).
* Subject has had a stable living arrangement at the time of screening and agrees to return to a similar living arrangement after discharge. This criterion is not meant to exclude subjects who have temporarily left a stable living arrangement (eg, due to psychosis). Such subjects remain eligible to participate in this study. Chronically homeless subjects should not be enrolled.
* Subject must agree to comply with all medication restrictions for the required length of time.

Exclusion criteria:

* 1. Subject answers "yes" to "Suicidal Ideation" Items 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS at or during the Screening period (ie, in the past one month) and/or Day 1 (ie, since last visit).

  2. Subject does not tolerate venipuncture or has poor venous access that would cause difficulty for administration of the radioisotope and for collecting blood samples.

  3. Subject is currently participating in, or has participated in, a study with an investigational or marketed compound or device within 3 months prior to signing the informed consent, or has participated in more than 2 studies of investigational compounds within 24 months prior to signing the informed consent.

  4. Subject has participated in a research and/or PET or radiological investigations with radiation exposure that, when combined with the dose from the present study, would exceed 10 mSv in addition to natural background radiation, in the previous 12 months.

  5. Subject has previously received SEP-363856.

  6. Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study:
  1. Clinically significant hematological (including deep vein thrombosis) or bleeding disorder, renal, metabolic, endocrine, pulmonary, gastrointestinal, urological, cardiovascular, hepatic, neurologic, or allergic disease (except for untreated, asymptomatic, seasonal allergies at time of dosing).
  2. Subject has a history of malignancy within 5 years prior to the Screening visit, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Subject has a pituitary tumor of any duration.
  3. Disorder or history of a condition, or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection) that may interfere with drug absorption, distribution, metabolism, excretion, gastrointestinal motility, or pH, or a history of clinically significant abnormality of the hepatic or renal system, or a history of malabsorption.
  4. Subject currently has or has had within the last 6 months a diagnosis of Alcohol or Substance Abuse Disorder (DSM-5 criteria). The only exceptions include caffeine or nicotine.
  5. Subject has a clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete the study as determined by the Investigator or a screening 12-lead ECG demonstrating any one of the following: heart rate > 100 beats per minute, QRS > 120 ms, QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms (males), QTcF > 470 ms (females), or PR > 220 ms.
  6. Subjects with known history of human immunodeficiency virus (HIV) seropositivity.
  7. Subject has a history of clinically significant hypotensive disorder, systolic blood pressure less than or equal to 80 mmHg or a diastolic blood pressure less than or equal to 40 mmHG at any measurement prior to dosing on Day 1, or any clinically significant symptoms associated with hypotension at any time during participation prior to dosing on day 1.

     7. Female subject who is pregnant or lactating.

     8 Subject has a presence or history of a medically diagnosed, clinically significant psychiatric disorder (including intellectual disability, major depressive disorder with psychosis, and bipolar disorder) other than schizophrenia (medically diagnosed schizoaffective disorder or schizophreniform disorder will be allowed).

     9. Subject tests positive for drugs of abuse at screening, however, a positive test for barbiturates, opiates, benzodiazepines or methadone may not result in exclusion of subjects if the Investigator determines that the positive test is as a result of prescription medicine(s). In the event a subject tests positive cannabinoids (tetrahydrocannabinol), the Investigator will evaluate the subject's ability to abstain from using this substance during the study. This information will be discussed with the Medical Monitor prior to study enrollment.

     10. Subject is at significant risk of harming him/herself or others according to the Investigator's judgment.

     11. Subject has attempted suicide within 6 months prior to screening.

     12. Subject is involuntarily hospitalized.

     13. Subject is judged in the opinion of the Investigator to be severely resistant to antipsychotic treatment defined as a failure to respond to 4 or more marketed antipsychotic agents, given at an adequate dose as per labeling and for an adequate duration (lifetime).

     14. Subject is receiving an antipsychotic medication at a dose above the maximum labeled dose (country-specific) dose at or during the 3 for less than 12 weeks prior to the PET scan at the screening visit

     15. Subject has received clozapine treatment within 120 days of planned PET scan at screening.

     16. Subject has received electroconvulsive therapy treatment within the 3 months prior to screening or is expected to require ECT during the study.

     17. Subject has a history of allergy or hypersensitivity to more than 2 distinct chemical classes of drug (eg, sulfonylureas and penicillins) allergic reaction to any medication or has a known or suspected sensitivity to any substance that is contained in the study drug formulation or to carbidopa or entacapone.

     18. Subject has any clinically significant abnormal laboratory values as determined by the Investigator (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, thyroid panel, and serum prolactin). (Note: abnormal findings of questionable significance will be discussed with the Medical Monitor prior to including subject).

     19. Subject demonstrates evidence of acute hepatitis, clinically significant chronic hepatitis, or evidence of clinically significant impaired hepatic function through clinical and laboratory evaluation. Note: Subjects with serum alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 3 times the upper limit of the reference ranges provided by the laboratory require retesting. If on retesting, the laboratory value remains ≥ 3 times the upper limit, the subject will be excluded.

     Note: subjects with serum alanine transaminase (ALT) or aspartate transaminase (AST) greater than or equal to 3 times the uper limit of the reference ranges provided by the laboratory require retesting. If on retesting, the laboratory value remains greater than or equal to 3 times the upper limit, the subject will be excluded.

     20. Subject has bilirubin greater than or equal to 1.5 x upper limit of normal (ULN) with the exception that isolated bilirubin greater than 1.5 x ULN is acceptable if bilirubin is fractioned and direct bilirubin less than 35% at screening.

     21. Subject has a serum blood urea nitrogen (BUN) or serum creatinine (Cr) value ≥ 1.5 times the upper limit of normal for the reference range.

     22. Subject has experienced significant blood loss (≥ 473 mL), has donated blood within 60 days prior to first dose of study drug, has donated plasma within 72 hours prior to the first dose of study drug or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.

     23. Subject consumes more than 300 mg of caffeine per day (5 cups of coffee or equivalent in caffeinated beverages).

     24. Subject has used disallowed prescription or disallowed nonprescription drugs, or dietary or herbal supplements as specified within the Concomitant Medications and Restrictions for at least 5 half-lives or 14 days prior to dosing, whichever is longer, or anticipates the need for any disallowed medication during their participation in this study (exception: female subjects who are taking oral, patch, or intrauterine device [IUD] hormonal contraceptives, or progestin implant or injection).

     25. Subject is a staff member or the relative of a staff member.

     26. Subject is in the opinion of the Investigator, unsuitable in any other way to participate in this study.

     27. Subject has contraindications to undergoing MRI/fMRI examination including, but not limited to claustrophobia, metal foreign bodies or implanted devices incompatible with the MRI/fMRI exposure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
  Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SEP-363856
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — SUBJECT WAS WITHDRAWN DUE TO SAFETY REASON | 1

BASELINE CHARACTERISTICS:
Arm/Group | SEP-363856
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Dopamine Synthesis Capacity at Week 2 Using 18F-DOPA.
Description: Dopamine synthesis capacity was assessed using 18 F-DOPA PET(positron emission tomography) scans that were performed before (baseline) and after (Week 2 [Day 14]) administration of SEP-363856 adjunctive to an antipsychotic medication. A repeated measures ANOVA(analysis of variance) analysis was conducted. The dependent variable was Dopamine Synthesis Capacity (Ki Values). The independent variables were Time and Striatal Subregion. The covariance matrix was unstructured for each subject's Time and Striatal Subregion.
Time Frame: baseline and week 2
Measure: Mean (Standard Deviation); unit: Kicer
Arm/Group | SEP-363856
Number analyzed (Participants) | 19
Kicer
  Whole Striatal Dopamine Synthesis Capacity | -0.0007 (0.00157)
  Limbic Striatal Dopamine Synthesis Capacity | -0.0008 (0.00118)
  Associative Striatal Dopamine Synthesis Capacity | -0.0006 (0.00158)
  Sensorimotor Striatal Dopamine Synthesis Capacity | -0.0008 (0.00207)
Statistical Analysis 1: Comparison: SEP-363856; To examine the primary outcome, the effects of SEP-363856 on the striatum, a repeated measures ANOVA model will be build using the baseline and on-treatment kicer values of each striatal subregion; Test type: Superiority; p = 0.0072, Repeated Measures ANOVA — A p-value of p<0.05 will be considered as significant

ADVERSE EVENTS:
Time Frame: Up to 36 days
Arm/Group | SEP-363856
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 19/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEP-363856 (N=22)
Vision blurred (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 4 (4)
Presyncope (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 14 (15)
Insomnia (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04038957/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT04038957/SAP_001.pdf